CLINICAL TRIAL: NCT06735534
Title: The ReMATCH Study is a Prospective, Single Arm, Open Label, Multi-center, Study Utilizing the FARAPULSE PFA System, Including the FARAWAVE and FARAPOINT PFA Catheters
Brief Title: Repeat Ablation of Persistent Atrial Fibrillation, Including Mitral Isthmus Catheter Ablation, With the FARAPULSE Pulsed Field Ablation System
Acronym: ReMATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF313
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Pulsed Field Ablation (PFA)); Pulmonary Vein Isolation; Recurrent Arrhythmia; cavo-tricuspid isthmus (CTI); CTI dependent flutter; Anti Arrhythmic Drugs (AAD); Atrial Flutter; Atrial Tachycardia; Atrial fibrillation; Electrical cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm Prospective (Other): Repeat Ablation of Persistent Atrial Fibrillation, including Mitral Isthmus Catheter Ablation, with the FARAPULSE Pulsed Field Ablation System.
  Interventions: Device: FARAPULSE™ Pulsed Field Ablation System

INTERVENTIONS:
Device: FARAPULSE™ Pulsed Field Ablation System — The FARAPULSE™ Pulsed Field Ablation System is indicated for the treatment of symptomatic atrial fibrillation.
  The FARAWAVE Catheter is indicated for the isolation of pulmonary veins and posterior wall in the treatment of drug-refractory, recurrent, symptomatic paroxysmal and persistent atrial fibrillation. The FARAWAVE Catheter is also indicated for the for the isolation of pulmonary veins and posterior wall in the treatment of persistent atrial fibrillation as an alternative to anti-arrhythmic drug (AAD) therapy as an initial rhythm control strategy.
  The FARAPOINT™ PFA Catheter is indicated for use as an adjunctive device for 1) the creation of an ablation line between the inferior vena cava and the tricuspid valve and/or 2) Mitral Isthmus, when the FARAWAVE Catheter is used in the endocardial treatment of persistent atrial fibrillation (episode duration no greater than 12 months).

SUMMARY:
The ReMATCH Study is a prospective, single arm, open label, multi-center, study utilizing the FARAPULSE PFA System, including the FARAWAVE and FARAPOINT PFA Catheters.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the safety and effectiveness of using the FARAWAVE™ and FARAPOINT™ pulsed field ablation (PFA) catheters for re-treatment of persistent atrial fibrillation (PersAF) after a failed initial procedure.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, or older if required by local law
* Single previous AF ablation procedure for Paroxysmal Atrial Fibrillation (PAF) or Persistent AF (PersAF)that minimally included pulmonary vein isolation that occurred within 5 years prior to enrollment.
* Documented (physician's note) diagnosis of PersAF either prior to the subject's Index Procedure OR development of PersAF after the Index Procedure.
* Documented evidence of AF recurrence at least 60 days after the subject's Index Procedure, captured by any regulatory cleared rhythm monitoring device.

OR

* If diagnosed with PersAF prior to the Index Procedure, documented recurrence of AF or atypical AFL at least 60 days after the Index Procedure, captured by any regulatory cleared rhythm monitoring device.
* Willing and capable of providing informed consent
* Willing and capable of participating in all follow-up assessments and testing associated with this clinical investigation at an approved clinical investigational center

Exclusion Criteria:

1. Atrial exclusions - Any of the following atrial conditions:

   1. Left atrial anteroposterior diameter ≥ 5.5 cm, or if LA diameter not available, non-indexed volume >100 ml (physician note or imaging)
   2. Current atrial myxoma
   3. Any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
   4. Current left atrial thrombus
2. Cardiovascular exclusions - Any of the following CV conditions:

   1. History of sustained ventricular tachycardia or any ventricular fibrillation
   2. AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
   3. Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, or implantable loop recorder, other than LUX-Dx.

      Prior interatrial baffle, atrial septal patch, atrial septal defect closure device, patent foramen ovale occluder, Amulet devices, or other left atrial appendage closure device if implanted within 90 days of enrollment
   4. Presence of any of the following:

      * Any prosthetic heart valve, ring or repair
      * Moderate to severe mitral valve stenosis
      * More than moderate mitral regurgitation (>3+)
      * Moderate to severe aortic stenosis
   5. Hypertrophic cardiomyopathy
   6. Any IVC filter, known inability to obtain vascular access or other contraindication to femoral access
   7. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
   8. Severe right ventricular dysfunction with documented echocardiography and/or hemodynamic data.
3. Any of the following conditions at baseline:

   1. Heart failure associated with NYHA Class III or IV
   2. Documented LVEF < 40% as documented within the previous 12 months
   3. Uncontrolled hypertension (SBP > 160 mmHg or DBP > 95 mmHg on two (2) BP measurements at baseline assessment not attributable to white coat syndrome per Investigator opinion
   4. Body Mass Index (BMI) >45.0
   5. CHA2DS2-VASc score ≥5
4. Any of the following events within 90 Days of the Consent Date:

   1. Coronary disease: Myocardial infarction (MI), unstable or Prinzmetal angina or coronary intervention within 90 days of consent or any documented history of severe non-revascularize coronary disease
   2. Cardiac surgery: Any cardiac surgery
   3. Heart failure hospitalization: Heart failure hospitalization
   4. Pericardium: Pericarditis or symptomatic pericardial effusion
   5. GI bleeding: Gastrointestinal bleeding
   6. Neurovascular event: Stroke, TIA, or intracranial bleeding
   7. Thromboembolism: Any active non-neurologic thrombus and/or thromboembolic event
   8. Carotid intervention: Carotid stenting or endarterectomy
   9. Diabetes: Uncontrolled diabetes mellitus or a recorded HgbA1c > 8.0%
5. Any of the following congenital conditions:

   1. Congenital heart disease: Congenital heart disease with any clinically significant residual anatomic or conduction abnormality
   2. Methemoglobinemia: History of known congenital methemoglobinemia
   3. G6PD deficiency: History of known G6PD deficiency
6. Any of the following conditions:

   1. Transplantation: Solid organ or hematologic transplant, or currently being evaluated for a transplant
   2. Diaphragmatic abnormality: Any prior history or current evidence of hemi-diaphragmatic paralysis or paresis
   3. Pulmonary: Severe lung disease, severe pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
   4. Renal: Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
   5. Malignancy: Active malignancy at enrolment (other than squamous cell carcinoma)
   6. Gastrointestinal: Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
   7. Infections: Active systemic infection
   8. Sleep apnea: Untreated diagnosed obstructive sleep apnea with apnea hypopnea index classification of severe (>30 pauses per hour)
   9. Medication use: Required use of phosphodiesterase inhibitors within 24 hours of the ablation procedure
   10. Nitroglycerin intolerance: Known allergic drug reaction to nitroglycerin (excluding hypotension)
   11. Hematologic condition: Known coagulopathy or bleeding disorder (e.g. von Willebrand disease, hemophilia)
   12. Contraindication to anticoagulation: Contraindication to, or unwillingness to use, systemic anticoagulation, or acceptable alternatives, pre-, intra- and post-procedure to achieve adequate anticoagulation.
   13. Pregnancy: Women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period
   14. General health conditions: Health conditions that in the investigator's medical opinion would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation.
   15. LUX-Dx ICM intolerance: Unwillingness to receive, or unable to tolerate, a subcutaneous, chronically inserted LUX-Dx ICM device
   16. Participation in another trial: Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility.
   17. Life expectancy: Predicted life expectancy less than three (3) years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint rate | 60 days
  The primary safety endpoint (PSE) is the proportion of Treatment subjects with one or more device or procedure-related Composite Serious Adverse Events (CSAEs) following the Repeat Ablation Procedure.
The primary effectiveness endpoint is the proportion of Treatment subjects with Acute Procedural Success. | 24 hours
  The proportion of Treatment Subjects with confirmed electrical block across all anatomical locations ablated with the investigational system only (Acute Procedural Success).

CONTACTS AND LOCATIONS:
Overall Officials: Moussa Mansour,, MD, Principal Investigator — Massachusetts General Hospital
Locations (25):
- United States (19):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arrhythmia Research Group-Research Facility, Jonesboro, Arkansas
  - University of Southern California Hospital, Los Angeles, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - HCA Florida Mercy Hospital, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - St. Luke's Boise Medical Center, Boise, Idaho
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Southcoast Physicians Group, Fall River, Massachusetts
  - Virtua Health Inc., Marlton, New Jersey
  - Bethesda North Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Trident Medical Center, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Australia (4):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Victorian Heart Hospital, Clayton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No